CLINICAL TRIAL: NCT07127445
Title: Metabolic and Epigenetic Impact of Concomitant Fatty Acid Amide Hydrolase Inhibitors and Oleoylethanolamide in a Novel Delivery
Brief Title: Metabolic and Epigenetic Impact of FAAH Inhibitors and OEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicole Stevens, PhD (Industry)
Responsible Party: Sponsor-Investigator, Nicole Stevens, PhD, Vice President, Clinical Research, dōTERRA International
Organization: dōTERRA International (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DO-124043-OEA
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Gene expression; Dietary supplement; OEA; Lavender essential oil; Ginger

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary supplement (Experimental): Participants take two capsules of the dietary supplement (one capsule in the morning and one in the evening) every day for 12 weeks.
  Interventions: Dietary Supplement: OEA supplement

INTERVENTIONS:
Dietary Supplement: OEA supplement — The supplement contains OEA, ginger extract, and lavender essential oil as its active ingredients.

SUMMARY:
The goal of this clinical trial is to learn whether a dietary supplement can affect gene expression and serum protein markers in healthy volunteers. The main questions it aims to answer are:

1. Does the supplement affect gene expression and protein markers as measured in blood?
2. How does daily ingestion of the supplement affect anthropometric measurements, including body mass index, waist circumference, blood pressure, and heart rate?
3. How does daily ingestion of the supplement affect subjective health parameters?
4. Is ingesting the supplement daily safe, as measured by laboratory tests and adverse events?

The supplement is made with oleoylethanolamide (OEA), ginger extract, and lavender essential oil.

Participants will:

* Take one supplement capsule in the morning and one in the evening every day for 12 weeks
* Attend three study visits in which they provide blood and urine samples, and undergo anthropometric measurements
* Complete surveys and subjective health assessments

DETAILED DESCRIPTION:
This open-label, repeated measures study will recruit healthy men and women to compare gene expression profile and serum protein markers before and after consumption of a dietary supplement for 12 weeks. Secondary outcomes include anthropometric measurements, vitals, and other subjective health assessments. Safety data (from blood sampling, urinalysis, and adverse events) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-64 years old
* BMI 25-30 inclusive (self-reported for screening, confirmed at first study visit)
* For purposes of blood collection and other in-person procedures:

  o Reside within driving distance of the study center or be willing to travel to the study center
* Willing and able to undergo three blood draws over 12 weeks
* Willing to wash out of all internally-consumed essential oils or botanical products for at least 2 weeks prior to starting the study, and willing to maintain the washout for the duration of the study (14 weeks).
* Willing and able to consume study product twice daily for about 12 weeks
* Willing to track consumption of study product
* Willing to keep diet, exercise, sleep habits, and current non-study supplement use the same throughout the study
* Willing to limit alcohol consumption to "social drinking" (typically no more than 3 drinks per day and 7 per week) during the study
* History of alcohol consumption limited to "social drinking" (typically no more than 3 drinks per day and 7 per week)
* Willing to avoid recreational drugs and smoking/vaping for the duration of the study (approximately 12 weeks)
* No metabolic disease (BMI>30, diagnosis and treatment of hypertension, diabetes, or dyslipidemia)
* No major diseases under treatment by doctor (Medical Reviewer's discretion)
* No pregnancy within the last 60 days or currently breastfeeding (females)
* No allergy to olive oil, lavender essential oil, ginger oleoresin/extract/essential oil, or OEA.
* No regular internal consumption of lavender essential oil, ginger oleoresin or extract, or OEA within the last 1 month (regularly is defined as dosing daily for more than 2 consecutive weeks, or dosing more than 2-3 times per week for 4 consecutive weeks)
* No evidence of medical condition, significant disease or disorder, medication, or surgery within the past 12 months that may, in the judgment of the medical provider, put the participant at risk or affect study results, procedures, or outcomes
* No recreational drug or smoking/vaping use in the past 1 month
* Not currently or previously participating in any other clinical trial within the last 30 calendar days

Exclusion Criteria:

* Failure to meet all inclusion criteria

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-19 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Gene expression | 6 weeks
  Gene expression analysis refers to a genome-wide quantification of methylation. EPIC850k array will be used for methylation analysis. This represents approximately 900,000 gene locations. The main feature performed is a differential methylation analysis to determine what has significantly changed from one time point to another. The changes will be evaluated before and after treatment with the study supplement for 6 weeks.
Hemoglobin A1C (HbA1c) (%) | 12 weeks
  Change in blood HbA1c value before and after 12 weeks of treatment with the study supplement.

SECONDARY OUTCOMES:
Comprehensive metabolic panel (CMP) | 12 weeks
  Panel used in safety assessment. Change in blood comprehensive metabolic panel values before and after 12 weeks of treatment with the study supplement, including:
  Albumin (g/dL) Blood urea nitrogen (BUN) (mg/dL) Creatinine (mg/dL) Alkaline phosphatase (U/L) Alanine transaminase (ALT) (U/L) Aspartate aminotransferase (AST) (U/L) Calcium (mg/dL) Carbon Dioxide (mmol/L) Chloride (mmol/L) Potassium (mmol/L) Sodium (mmol/L) Total bilirubin (mg/dL) Total protein (g/dL)
Complete blood count (CBC) | 12 weeks
  Panel used in safety assessment. Change in complete blood count values before and after 12 weeks of treatment with the study supplement, including:
  White blood cells (x10E3/uL) Red blood cells (x10E6/uL) Hemoglobin (g/dL) Hematocrit (%) Mean corpuscular volume (fL) Mean corpuscular hemoglobin (pg) Mean corpuscular hemoglobin concentration (g/dL) Red cell distribution width (%) Platelets (x10E3/uL) Neutrophils (%) Lymphocytes (%) Monocytes (%) Eosinophils (%) Basophils (%) Neutrophils (Absolute) (x10E3/uL) Lymphocytes (Absolute) (x10E3/uL) Monocytes (Absolute) (x10E3/uL) Basophils (Absolute) (x10E3/uL) Immature granulocytes (%) Immature granulocytes (Absolute) (x10E3/uL)
Generalized Anxiety Disorder-7 (GAD-7) scale | 12 weeks
  Validated, self-reported scale for the measurement of anxiety severity. The GAD-7 is a 7-item scale with total scores between 0 and 21. Higher scores indicate higher anxiety severity.
Leptin (ng/mL) | 12 weeks
  Change in blood leptin value before and after 12 weeks of treatment with the study supplement.
Apolipoprotein B (ApoB) (mg/dL) | 12 weeks
  Change in blood ApoB value before and after 12 weeks of treatment with the study supplement.
High sensitivity C-reactive protein (mg/dL) | 12 weeks
  Change in hsCRP (serum marker for inflammation and cardiac health) before and after treatment with the study supplement.
Patient Health Questionnaire (PHQ-8) scale | 12 weeks
  Validated, self-reported scale for the measurement of depression severity. The PHQ-8 is an 8-item scale with total scores between 0 and 12. Higher scores indicate higher depression severity.
Leeds Sleep Evaluation Questionnaire (LSEQ) scale | 12 weeks
  Validated, self-reported scale for the measurement of sleep quality. The LSEQ is a 10-item scale. Each item is scored 0 to 100. Higher scores indicate better sleep quality.
Body weight (kg) | 12 weeks
  Determine whether body weight (including body composition %) is affected by the consumption of the study product.
Lipid panel | 12 weeks
  Change in blood lipid panel values before and after 12 weeks of treatment with the study supplement, including:
  Total cholesterol (mg/dL) Triglycerides (mg/dL) High density lipoprotein (HDL) Cholesterol (mg/dL) Very Low density lipoprotein (VLDL) Cholesterol (mg/dL) Low density lipoprotein (LDL) Cholesterol (mg/dL)
Blood pressure (mmHg) | 12 weeks
  Determine whether blood pressure is affected by the consumption of the study product.
Heart rate (BPM) | 12 weeks
  Determine whether heart rate is affected by the consumption of the study product.
Waist circumference (cm) | 12 weeks
  Determine whether waist circumference is affected by the consumption of the study product.
Safety/tolerability | 12 weeks
  This study will monitor the occurrence and frequency of adverse events and safety, both through participant report and blood chemistry/hematology analyses.
Erythrocyte Sedimentation Rate (ESR) (mm/h) | 12 weeks
  Change in ESR (blood marker for inflammation) before and after treatment with the study supplement.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Stevens, PhD, Principal Investigator — doTERRA International
Locations (1):
- doTERRA International, Pleasant Grove, Utah, United States

IPD SHARING:
Plan to Share IPD: No